CLINICAL TRIAL: NCT03712826
Title: Identification by Cytometry by Mass of Predictive Immunological Profiles of Answer to Treatmentby Biotherapics for Patients With Crohn's Disease
Acronym: PICTURE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No inclusion
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL16_0811
Record Dates: First submitted 2018-08-16; First posted 2018-10-19 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Crohn Disease
Keywords: Crohn; immunological profile; ustekinumab; anti-TNF
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti TNF (Experimental): Crohn patient with antiTNF treatment
  Interventions: Drug: Anti-TNF Drug
- Ustekinumab (Experimental): Crohn disease with ustekinumab treatment
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Anti-TNF Drug — Crohn patient with antiTNF treatment
  Arms: anti TNF
Drug: Ustekinumab — Crohn disease with ustekinumab treatment
  Arms: Ustekinumab

SUMMARY:
Crohn disease is an inflammatory chronic disease of the bowel the complex physiopathology of which brings in immunological, genetic and environmental factors. At present, the appeal to biotherapics anti-TNFa (infliximab and adalimumab) or anti-IL-12/23 (ustekinumab) in MC represents a major therapeutic progress at the origin of a significant improvement of the symptoms, the healing of the intestinal hurts and the quality of life.

Considering the new immunological targets of these biotherapics, the investigators put the hypothesis that an immunological profile (impulsive person and\or tissular) specific of the patients with one MC is associated with the answer to biotherapics. So, before beginning the treatment the patients expressing strongly the pro-inflammatory cytokine TNFa, would more may be answering machines in anti-TNFa and those with whom the immunological profile is very marked towards the way Th1/Th17 would more may answer favorably the ustekinumab. The identification of immunological profiles capable of predicting before treatment the answer under biotherapics could establish in MC but also in other inflammatory diseases a major step forward to guide the coverage.

ELIGIBILITY:
Inclusion Criteria:

* Patient of more than 18 years old
* Patient presenting a MC before diagnosed according to the usual criteria
* Patient in relapse (score CDAI > 150) for at least 1 month
* requiring Patient a treatment by anti-TNF or ustekinumab according to the indications of the AMM
* Patient compatible with the realization of endoscopic digestive biopsies
* Patient having signed a consent of participation

Exclusion Criteria:

-· patient with Crohn disease with a CDAI score < 150 ·

* contraindication to anti-TNF and\or ustekinumab ·
* contraindication to the realization of an iléocoloscopie

  ·- Patient taking anti-inflammatory drugs or antibiotics ·
* Patient presenting complications of the type intestinal sub-occlusion, fistulas or abdominal abscesses ·
* Patient having a exclusive perianal disease or having
* pregnant Women ·
* Patients having been the object of a vast intestinal resection ·
* Patient with an ileostomy or a colostomy ·
* No consent of the patient ·
* patient under legal protection ·
* Subject participating in another research which need a period of exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
Immunological profile | Week 14
  Identify by cytometry of mass a predictive, blood and/or mucous immunological profile, of the answer at week 14 to a biotherapics by anti-TNFa or anti IL-12 / 23 at suffering patients of Crohn disease in relapse

SECONDARY OUTCOMES:
Mass cytometry dosage of immunological markers week 0-week 14 | Week 14
  Measurements of immunological markers by mass cytometry will be performed in the blood at baseline and at week 14 and in the gastrointestinal mucosa (endoscopic biopsies) only at baseline.
Clinical Remission at week 14 | Week 14
  Clinical remission will be defined as a reduction in the CDAI score ≤ 150 at week 14.
Dosage of inflammatory markers | week 14
  Assays for inflammatory blood (CRP) and fecal markers (fecal calprotectin) will be performed to predict the response to anti-TNFα or ustekinumab (anti IL-12/23) at inclusion and at week 14, with conventional methods used routinely.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Boschetti, MD, Principal Investigator — Hospices Civils de Lyon